CLINICAL TRIAL: NCT03996018
Title: T-cell Responses to Concurrent HIV and Herpesvirus Infections
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TORCH
Record Dates: First submitted 2019-05-29; First posted 2019-06-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: HIV; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1(HIV Uninfected): Participant is HIV negative per antibody screen conducted on premises and participant is enrolled on HPTN 083 study
  Interventions: Other: T-cell lymphocyte responses
- group 2 (HIV Infected): Participant has initiated ART therapy as a patient at St Jude Children's Research Hospital, newly diagnosed HIV and prolonged HIV
  Interventions: Other: T-cell lymphocyte responses

INTERVENTIONS:
Other: T-cell lymphocyte responses — T-cell lymphocyte responses to human immunodeficiency virus (HIV) with and without concomitant herpesvirus infections (specifically, the persistence of HIV-specific human CD8 T-cells in the context of antiretroviral therapy (ART).

SUMMARY:
This is a research study in which we are trying to discover new information about how HIV and herpes viruses interact with the immune system. The goal of the study is to learn more about how T-cells in your immune system respond to and fight off long-term (chronic) viruses, in order to improve medical care in the future.

DETAILED DESCRIPTION:
HIV-uninfected & HIV-infected participants who enroll on this study will be asked to provide blood samples for 18 months. These samples will be used to assess T-cell responses and presence of herpesvirus(es).

Primary Objective

Characterize phenotypic and functional features, including TCR repertoires of HIV-specific CD8 T-cell responses and exhaustion in HIV-positive humans with and without concomitant herpesvirus infections.

ELIGIBILITY:
Inclusion Criteria:

* Criteria • Participant is greater than or equal to 18 years of age.

Group 1 (HIV Uninfected) Only

* Participant is HIV negative per antibody screen conducted on premises
* Participant is enrolled on HPTN 083 study (receiving HIV-PrEP) (see Recruitment and Screening).

Group 2 (HIV Infected) Only

* Participant has initiated ART therapy as a patient at St Jude Children's Research Hospital

  *Note: participants will be allowed to continue on study and have data analyzed regardless of presence of detectable HIV or CD4+ counts.

  a) Newly diagnosed HIV
* Participant is HIV-1 positive per medical record documentation or positive antibody screen conducted on premises, with initial diagnosis within 90 days prior to enrollment

  b) Prolonged HIV
* Participant is HIV-1 positive per medical record documentation or positive antibody screen conducted on premises, with initial diagnosis more than 365 days prior to enrollment

Exclusion Criteria:

* Participant is unable or unwilling to provide informed consent.
* If female of child bearing potential, participant has a positive urine pregnancy test at screening. Note: if participant becomes pregnant while on study, they may not continue on study.
* Concurrent enrollment on a research study or receiving treatment for concurrent medical diagnosis with any of the following interventions which may impact study outcomes: high dose or prolonged steroids, chemotherapy to treat malignancy, radiation therapy, biologic pharmaceutical treatments that induce immunosuppression.
* If in the opinion of the investigator, participation in the blood draw would endanger the health of the participant.
* Participant is enrolled in other clinical trials that include any blood sampling such that the cumulative blood draws would exceed that established as constituting minimal risk (e.g., more than 550 ml in an 8 week period with collection more frequently than 2 times per week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with HIV who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
HIV-1 specific TCR repertoire: Change in Simpson's diversity index over time | 0, 6, 12 and 18 months (+/- 30 days for all time points after 0).
  using separated PBMCs, HIV-1 specific T-cells will be labeled with major histocompatibility complex (MHC) I tetramers previously described to be specific for HIV-1 [14-18]. Labeled cells will be subjected to flow cytometry for identity confirmation via established antibody cell marker staining, counting and sorting into single cells. The TCR genes of the individually sorted HIV-1 tetramer positive T-cells will then be sequenced, establishing a repertoire of TCR sequences. Diversities of the TCR gene repertoires obtained from each study group will be assessed using the established algorithm for Simpson's diversity index [9].

SECONDARY OUTCOMES:
Herpesvirus specific TCR repertoire: Change in Simpson's diversity index | 0, 6, 12 and 18 months (+/- 30 days for all time points after 0).
  process as described above, with use of newly identified and previously published herpesvirus specific MHC I tetramers, including those for HSV-1, HSV-2, EBV and CMV, [19-25]. Comparisons of TCR repertoires will be made between newly acquired and latent herpesvirus infections. Diversities of the TCR gene repertoires obtained from each study group will be assessed using the established algorithm for Simpson's diversity index [9].
T-Cell exhaustion: binary value (Exhausted/not exhausted) | 0, 6, 12 and 18 months (+/- 30 days for all time points after 0
  Intracellular and cell surface proteins will be assessed to determine if T-cells that have entered the exhaustion pathway. These markers include, but are not limited to, PD-1, Tim3, Tcf7, Tbet, and Tox. Marker expression will be measured at the transcript or protein level [1, 2]; T-cells will be concomitantly labeled/detected with T-cell specific markers and HIV-1 MHC I tetramers to confirm identity. Using this information, a binary value of "exhausted' or "not exhausted" will be assigned.
HIV control: HIV viral load | 0, 6, 12 and 18 months (+/- 30 days for all time points after 0
  presence (or lack of) of HIV infection will be determined by HIV antigen/antibody testing. Control will be assessed by CD4+ T-cell counts, HIV viral titers, infections acquired likely due to immunodeficiency. The main outcome measure will be viral load. HIV related laboratory results including HIV screen, viral titers, T-cell counts will all be disclosed to patients as per standard of care.
Presence of herpesvirus infections: IgM and IgG levels | 0, 6, 12 and 18 months (+/- 30 days for all time points after 0
  at first visit, all patients will have IgM and IgG levels in the clinical laboratory for each named virus to establish presence of chronic vs. newly acquired herpesvirus infections. At each visit all patients will have serological testing via HSV-1, HSV-2, CMV, EBV and specific IgG direct antibody detection with quantitative enzymatic immune assay (EIA). Patients with active mucosal (oral or genital) or skin lesions consistent with primary or secondary HSV infections will be swabbed and sent for PCR and/or direct fluorescence antibody assay (DFA) in the clinical laboratory. Control will be assessed by quantitative EIA results and frequency of herpesvirus specific symptoms of flare (acute or reactivated infections).
HLA typing | baseline
  peripheral blood mononuclear cells (PBMCs) will be separated from patient's whole blood specimens. DNA will be extracted and specific HLA loci will be amplified using PCR, and yielded products will be sequenced. This will guide appropriate use of TCR tetramers.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Green, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols